CLINICAL TRIAL: NCT04062123
Title: Modulation of Memory and Conditioning by Pain During Sedation With Anesthetics
Brief Title: Memory & Conditioning Under Anesthesia
Acronym: MCA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Keith M Vogt (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor-Investigator, Keith M Vogt, Associate Professor of Anesthesiology & Perioperative Medicine and Bioengineering, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY19030183; R35GM146822 (NIH)
Record Dates: First submitted 2019-07-11; First posted 2019-08-20 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Anesthesia; Pain
Keywords: propofol; dexmedetomidine; fentanyl; functional MRI; electric nerve stimulation; sedation; functional connectivity
MeSH Terms: conditions — Pain | interventions — Dexmedetomidine; Propofol; Fentanyl; Transcutaneous Electric Nerve Stimulation; Sodium Chloride; Fluid Therapy

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, within-subject, crossover between no-drug and assigned drug (in randomized order)
Who Masked: Participant
Masking Description: single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Dexmedetomidine (Experimental): Subjects in this group will receive dexmedetomidine during the drug portion of the experiment.
  Interventions: Drug: Dexmedetomidine; Device: Peripheral Nerve Stimulation; Drug: Placebo
- Propofol (Experimental): Subjects in this group will receive propofol during the drug portion of the experiment.
  Interventions: Drug: Propofol; Device: Peripheral Nerve Stimulation; Drug: Placebo
- Fentanyl (Experimental): Subjects in this group will receive fentanyl during the drug portion of the experiment.
  Interventions: Drug: Fentanyl; Device: Peripheral Nerve Stimulation; Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Subjects in this group will receive a intravenous infusion of this drug, during a portion of the study. Dose will be targeted to a brain effect site concentration of 0.15 ng/ml, using pharmacokinetic modelling within the STANPUMP algorithm that accounts for subject's age, gender, height, & weight.
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Propofol — Subjects in this group will receive a intravenous infusion of this drug, during a portion of the study. Dose will be targeted to a brain effect site concentration of 0.7 mcg/ml, using pharmacokinetic modelling within the STANPUMP algorithm that accounts for subject's age, gender, height, & weight.
  Other Names: Diprivan
  Arms: Propofol
Drug: Fentanyl — Subjects in this group will receive a intravenous infusion of this drug, during a portion of the study. Dose will be targeted to a brain effect site concentration of 0.9 ng/ml, using pharmacokinetic modelling within the STANPUMP algorithm that accounts for subject's age, gender, height, & weight.
  Other Names: fentanyl citrate
  Arms: Fentanyl
Device: Peripheral Nerve Stimulation — Experimental acute pain stimulus will be delivered using a nerve stimulator. These painful shocks will be paired randomly with some of the experimental cues.
  Other Names: Electric Nerve Stimulation
Drug: Placebo — Crystalloid IV solution will be infused, with no active drug.
  Other Names: saline, IV fluid

SUMMARY:
The purpose of this study is to determine the effects of pain on long-term memory and conditioned physiologic responses in the presence and absence of distinct intravenous anesthetics. Functional magnetic resonance imaging will be used to identify the neural correlates of these phenomena The study will occur over 5 visits and involves no long-term follow up.

DETAILED DESCRIPTION:
Purpose: Sedative-hypnotic and analgesic agents (termed "anesthetics") are routinely used during medical procedures to prevent or ease suffering, suppressing the conscious experience of pain and its encoding into memory. While overt awareness under general anesthesia is a rare clinical event, implicit memory may still form. Further, at sub-hypnotic anesthetic doses, animals show enhanced fear conditioning and humans may have enhanced amygdala activity. This motivates the investigator's study, as poorly-contextualized aversive memories are theorized to initiate anxiety-spectrum disorders, which may explain the high incidence of post-traumatic stress disorder after anesthetic awareness.

Objective: How anesthetics facilitate or inhibit poorly-contextualized aversive memories is incompletely understood, with little mechanistic work done in human subjects. Thus, there is a critical need to understand how anesthetics modulate the memory and threat response systems during painful stimulation. The overall scientific objective is to determine the memory-modulating effects of propofol, dexmedetomidine, and fentanyl in the context of periodic painful stimulation.

Aim 1: Determine how behavioral and physiologic measures of memory are modulated by pain and the individual effects of three pharmacologically distinct drugs: propofol, dexmedetomidine, and fentanyl. Hypotheses: Based on previous results, 1a) explicit memory will be significantly reduced by propofol and dexmedetomidine, but only modestly by fentanyl. Consistent with my preliminary data, 1b) priming effects will be seen for pain-paired words under all drugs. Electrodermal activity changes still occur with opioids and propofol, thus 1c) pain-related physiologic responses will persist with these two drugs but be blunted by the anti-adrenergic effect of dexmedetomidine.

Aim 2: Determine the brain structures differentially engaged in memory encoding under pain and drug conditions. Task-related functional magnetic resonance imaging (MRI) activity for behavioral measures of explicit or implicit memory will be determined, comparing pain-paired vs non-pain items across drug and no-drug datasets. Functional connectivity (FC) MRI (fcMRI) will be compared between task and drug conditions. The entire brain will be explored, but predictions for key structures follow. Hypotheses: 2a) Hippocampal activity, will be blunted by propofol and dexmedetomidine, while fentanyl will have minimal effect. 2b) Amygdala activity, responsible for physiologic responses, will parallel the predictions in 1c across drug and pain conditions. 2c) Insula activity will be greater for pain-paired items, and this will be attenuated by fentanyl > dexmedetomidine > propofol, corresponding to their anticipated analgesic effect. 2d) Pain has been shown to affect fcMRI during a cognitive task, and thus FC between the key regions in 2a-c will be reduced by all three drugs, in characteristic patterns.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age 18-39, who are native English speakers with at least a high school education
* have normal hearing and memory
* be of normal body-weight
* be generally healthy (free from significant chronic disease)
* have none of the specific exclusion criteria
* have a valid email address and valid phone number throughout the study
* anticipate ability to participate in all visits required for the phase of the study in which they are enrolled

Exclusion Criteria:

* Pregnancy
* Body mass index > 35 (obese) or < 18 (underweight)
* Use of psychotropic medications, including anti-epileptics, anti-psychotics, anxiolytics, anti-depressants, stimulants, sleep-aids, anti-histamines, or analgesics
* History of adverse reaction to OR abuse of: dexmedetomidine (Precedex), propofol (Diprivan) or the opioids class of medications (fentanyl, morphine, hydromorphone, etc)
* History of clinically significant memory or hearing loss
* History of obstructive sleep apnea
* History of neurologic or psychiatric disease, including benign tremor
* History of significant cardiac disease, including high blood pressure or arrhythmia
* History of significant pulmonary disease
* History of diabetes or neuropathy
* History of chronic pain, or other pain processing disorder
* Have an implanted medical electronic device
* Have indwelling or implanted metal in their body that is not MRI-compatible
* Have claustrophobia
* Have a history of drug abuse

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith M Vogt, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Propofol: Subjects in this group received propofol during the drug portion of the experiment.
- Dexmedetomidine: Subjects in this group received dexmedetomidine during the drug portion of the experiment.
- Fentanyl: Subjects in this group received fentanyl during the drug portion of the experiment.
Period: Overall Study
Arm/Group | Propofol | Dexmedetomidine | Fentanyl
Started | 30 | 29 | 33
Completed | 30 | 28 (One subject did not complete the study) | 33
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Propofol: Subjects in this group received intravenous propofol, during a portion of the study. Dose was targeted to an effect site concentration of 1.0 mcg/ml, using pharmacokinetic modelling that accounts for subject's age, gender, height, & weight.
- Dexmedetomidine: Subjects in this group received intravenous dexmedetomidine, during a portion of the study. Dose was targeted to an effect site concentration of 0.15 ng/ml, using pharmacokinetic modelling that accounts for subject's age, gender, height, & weight.
- Fentanyl: Subjects in this group received intravenous fentanyl, during a portion of the study. Dose was targeted to a brain effect site concentration of 0.9 ng/ml, using pharmacokinetic modelling that accounts for subject's age, gender, height, & weight.
- Total: Total of all reporting groups
Arm/Group | Propofol | Dexmedetomidine | Fentanyl | Total
Number analyzed (Participants) | 30 | 29 | 33 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.0 (6.2) | 25.6 (6.5) | 23.9 (5.0) | 24.8 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 16 | 45
  Male | 16 | 14 | 17 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 3 | 7
  Not Hispanic or Latino | 22 | 22 | 27 | 71
  Unknown or Not Reported | 7 | 4 | 3 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 6 | 8 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 3 | 3
  White | 18 | 17 | 15 | 50
  More than one race | 0 | 2 | 4 | 6
  Unknown or Not Reported | 7 | 4 | 3 | 14
Region of Enrollment [Number; unit: participants]
  United States | 30 | 29 | 33 | 92

OUTCOME MEASURES:

1. Primary Outcome: Explicit Memory Performance
Description: Recognition memory testing, using the Remember-Know procedure, in which subjects indicate whether they recognize previously experienced experimental items among novel items (not previously in the experiment). This allows calculation of interdependent measures of recollection & familiarity using the signal detection statistic, d'. d' is calculated as the cumulative Gaussian distribution of false positive responses subtracted from the cumulative Gaussian distribution of correctly identified previously-experienced items. d' is on a (theoretically infinite) scale of standard deviation units, with negative values representing performance worse than chance guessing and positive values representing stand deviations of performance above chance.
Time Frame: 24-hrs post-experiment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Placebo Control: Data obtained from subjects across all three drug groups, during portion of experiment receiving no drug.
- Propofol: Data from subjects assigned to propofol group, from experimental session in which they were under a steady-state effect site concentration of propofol of 1.0 mcg/ml.
- Dexmedetomidine: Data from subjects assigned to dexmedetomidine group, from experimental session in which they were under a steady-state effect site concentration of dexmedetomidine of 0.15 ng/ml.
- Fentanyl: Data from subjects assigned to fentanyl group, from experimental session in which they were under a steady-state effect site concentration of fentanyl of 0.9 ng/ml.
Arm/Group | Placebo Control | Propofol | Dexmedetomidine | Fentanyl
Number analyzed (Participants) | 92 | 30 | 29 | 33
units on a scale | 1.16 [0.97 to 1.34] | .51 [0.182 to 0.842] | 1.04 [0.73 to 1.35] | .98 [0.68 to 1.28]

2. Secondary Outcome: Brain Activation in the Hippocampus for Successful Memory Formation: Placebo Condition Minus Drug Condition
Description: The Z-score is calculated by linear regression of the task timing against the MRI signal time-course (MRI data is in arbitrary units with no maximum or minimum) at each voxel (single data point in brain). The outcome is listed for the hippocampus, but similar scores are calculated throughout the brain. Z-score of 0 indicates no task-related changes. Z-scores further from zero indicate a larger difference in brain activity, with positive values indicating decreases under the drug condition, while negative Z-scores indicate increases under drug, compared to control. This outcome is reported as a number, as it is calculated using all the data across subjects combined into one statistical measure for the overall strength of difference in MRI signal change between two groups of data. Dispersion measures cannot be calculated for the summary Z-score.
Time Frame: Immediately after each experimental item
Measure: Number; unit: Z-score for difference
Arm/Group | Propofol | Dexmedetomidine | Fentanyl
Number analyzed (Participants) | 30 | 29 | 33
Z-score for difference | 3.8 | -4.9 | -5.0

3. Secondary Outcome: Heart Rate Response
Description: Heart rate changes (measured by electrocardiogram, EKG) were planned to be determined following experimental stimuli that delivered as part of the experiment. A 1-6 second window of physiologic data will be analyzed for changes in the peak of the EKG response (R-wave), allowing calculation of instantaneous heart rate. Increases in heart rate are well-known to correlate to sympathetic nervous system activity increases.
Time Frame: Immediately after each experimental item
Population: Acquisition of EKG data was not possible in the scanner, due to interference from the magnetic field. This is why the outcome cannot be reported.
Arm/Group | Propofol | Dexmedetomidine | Fentanyl
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Skin Response
Description: Electrodermal activity (galvanic skin) response was planned to be determined following experimental stimuli that delivered as part of the experiment. A 1-6 second window of physiologic data will be analyzed for changes in electrodermal activity, measured from the palm of subjects' hand. this well-established measure indicates sweat gland activity and is correlated to sympathetic nervous system activity increases.
Time Frame: Immediately after each experimental item
Population: Acquisition of skin conductance data was not possible in the scanner, due to interference from the magnetic field. This is why the outcome cannot be reported.
Arm/Group | Propofol | Dexmedetomidine | Fentanyl
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout the entire study period, at 5 study visits taking place over up to 3 months.
Arm/Group | Propofol | Dexmedetomidine | Fentanyl
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/29 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29 | 0/33
Other Adverse Events (participants affected / at risk) | 0/30 | 0/29 | 2/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propofol (N=30) | Dexmedetomidine (N=29) | Fentanyl (N=33)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/23/NCT04062123/Prot_001.pdf
  • Statistical Analysis Plan (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/23/NCT04062123/SAP_002.pdf
  • Informed Consent Form (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/23/NCT04062123/ICF_000.pdf